CLINICAL TRIAL: NCT04672291
Title: A Phase I-Ib, Double-blinded, Randomized Repeated Dose Single Center, Safety and Immunogenicity Study of Nasal Poly-ICLC (Hiltonol®) in Healthy COVID-19 Vaccinated Adults
Brief Title: Nasal Poly-ICLC (Hiltonol®) in Healthy COVID-19 Vaccinated Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncovir, Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ONV2020-003
Record Dates: First submitted 2020-10-05; First posted 2020-12-17 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: COVID - 19
Keywords: SARS CoV-2; COVID; Prevention; Poly-ICLC; Viral Infection
MeSH Terms: conditions — COVID-19; Virus Diseases | interventions — poly ICLC; Safety

STUDY DESIGN:
Intervention Model Description: Intranasal Poly-ICLC (Hiltonol®) or Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study consists of 2 treatment groups. Study subjects will be assigned by chance to a treatment group. Group 1 receives the study drug; group 2 receives the placebo. Neither the study subject or the study team will know the group assignments. There will be a 4 out 5 chance of receiving the study drug and 1 out 5 chance of receiving the placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Cohort (Experimental): A randomized (4:1) initial safety cohort of 13 patients will receive 2 cycles of drug (N=10) or placebo (N=3)
  Interventions: Drug: Poly-ICLC (Hiltonol®) or Placebo
- Expansion Cohort (Experimental): A randomized (4:1) expansion cohort will receive 3 cycles of drug (N=24) or placebo (N=6). A total of 30 patients will be accrued.
  Interventions: Drug: Poly-ICLC (Hiltonol®) or Placebo

INTERVENTIONS:
Drug: Poly-ICLC (Hiltonol®) or Placebo — The safety cohort (Cohort A) consists of 13 patients who will be randomized to receive 2 cycles of the study drug (N10) or 2 placebo cycles (N3).
  Other Names: Safety
  Arms: Safety Cohort
Drug: Poly-ICLC (Hiltonol®) or Placebo — The expansion cohort will receive 3 cycles of therapy. A total of 30 patients will be accrued and randomized 4:1 to receive drug (N=24) or placebo (N=6).
  Other Names: Expansion
  Arms: Expansion Cohort

SUMMARY:
This is a randomized (4:1) Phase 1 b safety trial in adults who have completed their full COVID-19 vaccination schedule at least 30 days prior to study entry.

DETAILED DESCRIPTION:
An initial cohort of 13 participants will receive 2 cycles of drug or placebo per the schedule below under carefully monitored conditions, including examinations to observe and document administration site reaction following consecutive administration cycles of the drug. 10 participants will receive drug and 3 will receive placebo. The safety stopping rule is to implement an enrollment pause if 2 dose limiting toxicity (DLT, see section 5.1) out of the first six or 3 DLTs out of the first 10 participants receiving drug are observed in either cycle 1 or cycle 2. The independent DSMB will conduct a review of the safety data to determine the relatedness of the DLTs to the drug exposure and provide a recommendation to continue. Thus, if safety events are determined to be not (or unlikely) related to drug exposure the trial may resume. The independent DSMB will review safety and tolerance data before the study can continue.

If at most 2 DLTs out of the 10 participants receiving drug are observed, then a Phase Ib expansion cohort will open. The expansion cohort will receive 3 cycles of therapy. A total of 30 participants will be accrued and randomized 4:1 to receive drug (N=24) or placebo (N=6). There will be extensive assessment of toxicity and an early stopping rule to implement an enrollment pause and independent DSMB review of safety data to determine relatedness to drug exposure for recommendation of trial continuation, will be employed as above. Safety and tolerability will be the primary endpoint but secondary endpoints include changes in immunological parameters.

ELIGIBILITY:
Inclusion Criteria for Enrollment

1. Phase I Cohort A: Subjects must be between 18 and 69 years of age. Phase 1b Cohort B: Subjects must be 18 years of age or older. In order to mitigate risk, no participants over age 70 will be recruited in Cohort A.
2. Asymptomatic; defined by experiencing none of the symptoms identified in the Symptom Questionnaire

   1. fever
   2. cough
   3. dyspnea
   4. fatigue
   5. muscle or joint pain
   6. sore throat
   7. stuffy or runny nose
   8. nausea/vomiting
   9. headache
   10. confusion
   11. diarrhea
   12. loss of smell or taste
3. Nasopharyngeal swab for COVID-19 at screening with negative diagnosis of SARS-CoV-2
4. Willing and able to provide blood, nasopharyngeal swab, and nasal mononuclear samples
5. Healthy individuals fully vaccinated with a COVID-19 vaccine and who have had their last dose of COVID-19 vaccination at least 30 days prior to study entry. Healthy individuals vaccinated with a COVID-19 booster shot are eligible for enrollment. The vaccination dates of the doses, and specific vaccine received will be recorded.
6. Able to provide informed consent
7. Female participants of childbearing potential and male participants with partners of childbearing potential must agree to use adequate methods of contraception (described below) during the study treatment and through 90 days after the last dose of study medication. Female participants of childbearing potential are all those except participants who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal
8. Acceptable Hematologic, renal and liver functions as follows:

1. Absolute neutrophil count > 1000/mcL 2. Platelets > 50,000/mcL 3. Hemoglobin >9 g/dL 4. Serum Creatinine ≤ 2.5 mg/dl 5. Liver Function:

* Total bilirubin ≤1.5 mg/dl
* AST ≤ 2.0 mg/dl (≤120 IU or 3x ULN)

Exclusion Criteria

1. Individuals not yet fully vaccinated with a COVID-19 vaccine.
2. Receipt of any blood product in past 120 days
3. Allergic rhinitis, chronic sinusitis, or other nasal inflammatory disease that requires daily intranasal or oral medication
4. Chronic medical problems that require daily nasal administration of medication
5. Prior nasal or sinus surgery including trans nasal approaches to brain
6. Chronic pulmonary conditions including severe asthma, COPD, or chronic bronchitis
7. Autoimmune hepatitis, decompensated liver disease, cardiac ischemia, congestive heart failure, cardiac arrhythmia, neutropenia, thrombocytopenia, severe renal insufficiency
8. Psychiatric or cognitive illness or recreational drug/alcohol use that in the opinion of the principal investigator, would affect participant safety and/or compliance
9. Symptoms consistent with COVID-19 infection (fevers, acute onset cough, shortness of breath) at time of screening
10. Nucleic acid testing evidence of COVID-19 infection at time of screening
11. Participants must not be pregnant or nursing due to the unknown potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
12. Has a diagnosis of primary immunodeficiency
13. Has uncontrolled hypertension that in the opinion of the principal investigator poses unacceptable risk.
14. Has active autoimmune disease that has required systemic treatment in the past 1 year

    1. (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs)
    2. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is acceptable
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating Investigator
16. Principle investigator believes that for one or multiple reasons the participant will be unable to comply with all study visits, or if they believe the trial is not clinically in the best interest of the participant
17. Documented allergic or hypersensitivity response to any protein therapeutics (e.g., recombinant proteins, vaccines, intravenous immune globulins, monoclonal antibodies, receptor traps)
18. Active, untreated tuberculosis

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of nasally administered Poly-ICLC (Hiltonol®) in healthy adults. | 91 days
  Safety will be measured and tabulated by the number (percent) of participants who experience DLTs (grade 3/4 adverse events) from the start of therapy through the end of the follow up period (day 91), according to DAIDS.

SECONDARY OUTCOMES:
Assess the response of the body to the study drug (pharmacodynamics) | 91 days
  Characterize the pharmacodynamics of the local and systemic innate immune response to repeated doses of intranasal Poly-ICLC (Hiltonol®) by investigating the effects on nasal mononuclear cells and systemic inflammatory markers

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Salazar, MD, Study Director — Sponsor GmbH
Locations (1):
- Health Research Innovation Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams JG, Walls RM. Supporting the Health Care Workforce During the COVID-19 Global Epidemic. JAMA. 2020 Apr 21;323(15):1439-1440. doi: 10.1001/jama.2020.3972. No abstract available. PMID 32163102
- [Result] Antonelli LR, Gigliotti Rothfuchs A, Goncalves R, Roffe E, Cheever AW, Bafica A, Salazar AM, Feng CG, Sher A. Intranasal Poly-IC treatment exacerbates tuberculosis in mice through the pulmonary recruitment of a pathogen-permissive monocyte/macrophage population. J Clin Invest. 2010 May;120(5):1674-82. doi: 10.1172/JCI40817. Epub 2010 Apr 12. PMID 20389020
- [Result] Balan S, Arnold-Schrauf C, Abbas A, Couespel N, Savoret J, Imperatore F, Villani AC, Vu Manh TP, Bhardwaj N, Dalod M. Large-Scale Human Dendritic Cell Differentiation Revealing Notch-Dependent Lineage Bifurcation and Heterogeneity. Cell Rep. 2018 Aug 14;24(7):1902-1915.e6. doi: 10.1016/j.celrep.2018.07.033. PMID 30110645
- [Result] Benveniste EN, Qin H. Type I interferons as anti-inflammatory mediators. Sci STKE. 2007 Dec 11;2007(416):pe70. doi: 10.1126/stke.4162007pe70. PMID 18073382
- [Result] Boukhvalova MS, Sotomayor TB, Point RC, Pletneva LM, Prince GA, Blanco JC. Activation of interferon response through toll-like receptor 3 impacts viral pathogenesis and pulmonary toll-like receptor expression during respiratory syncytial virus and influenza infections in the cotton rat Sigmodon hispidus model. J Interferon Cytokine Res. 2010 Apr;30(4):229-42. doi: 10.1089/jir.2009.0025. PMID 20038196
- [Result] CDC COVID-19 Response Team. Characteristics of Health Care Personnel with COVID-19 - United States, February 12-April 9, 2020. MMWR Morb Mortal Wkly Rep. 2020 Apr 17;69(15):477-481. doi: 10.15585/mmwr.mm6915e6. PMID 32298247
- [Result] Caskey M, Lefebvre F, Filali-Mouhim A, Cameron MJ, Goulet JP, Haddad EK, Breton G, Trumpfheller C, Pollak S, Shimeliovich I, Duque-Alarcon A, Pan L, Nelkenbaum A, Salazar AM, Schlesinger SJ, Steinman RM, Sekaly RP. Synthetic double-stranded RNA induces innate immune responses similar to a live viral vaccine in humans. J Exp Med. 2011 Nov 21;208(12):2357-66. doi: 10.1084/jem.20111171. Epub 2011 Nov 7. PMID 22065672
- [Result] Christopher ME, Wong JP. Use of TLR3 receptor agaonists against respiratory viral infections. Anti-inflammatory & Anti-Allergy Agents in Medicinal Chemistry. 2011;10:327-38.
- [Result] Flynn BJ, Kastenmuller K, Wille-Reece U, Tomaras GD, Alam M, Lindsay RW, Salazar AM, Perdiguero B, Gomez CE, Wagner R, Esteban M, Park CG, Trumpfheller C, Keler T, Pantaleo G, Steinman RM, Seder R. Immunization with HIV Gag targeted to dendritic cells followed by recombinant New York vaccinia virus induces robust T-cell immunity in nonhuman primates. Proc Natl Acad Sci U S A. 2011 Apr 26;108(17):7131-6. doi: 10.1073/pnas.1103869108. Epub 2011 Apr 5. PMID 21467219
- [Result] Guerrero-Plata A, Baron S, Poast JS, Adegboyega PA, Casola A, Garofalo RP. Activity and regulation of alpha interferon in respiratory syncytial virus and human metapneumovirus experimental infections. J Virol. 2005 Aug;79(16):10190-9. doi: 10.1128/JVI.79.16.10190-10199.2005. PMID 16051812
- [Result] Hill DA, Baron S, Perkins JC, Worthington M, Van Kirk JE, Mills J, Kapikian AZ, Chanock RM. Evaluation of an interferon inducer in viral respiratory disease. JAMA. 1972 Feb 28;219(9):1179-84. No abstract available. PMID 4334380
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Kato H, Takeuchi O, Sato S, Yoneyama M, Yamamoto M, Matsui K, Uematsu S, Jung A, Kawai T, Ishii KJ, Yamaguchi O, Otsu K, Tsujimura T, Koh CS, Reis e Sousa C, Matsuura Y, Fujita T, Akira S. Differential roles of MDA5 and RIG-I helicases in the recognition of RNA viruses. Nature. 2006 May 4;441(7089):101-5. doi: 10.1038/nature04734. Epub 2006 Apr 9. PMID 16625202
- [Result] Kende M, Paragas J, Salazar AM. The efficacy of poly-ICLC against Ebola-Zaire virus (EBOV) infection in mice and cynomolgus monkeys. Antiviral Res. 2019 Mar;163:179-184. doi: 10.1016/j.antiviral.2018.12.020. Epub 2019 Jan 3. PMID 30611774
- [Result] Kindler E, Gil-Cruz C, Spanier J, Li Y, Wilhelm J, Rabouw HH, Zust R, Hwang M, V'kovski P, Stalder H, Marti S, Habjan M, Cervantes-Barragan L, Elliot R, Karl N, Gaughan C, van Kuppeveld FJ, Silverman RH, Keller M, Ludewig B, Bergmann CC, Ziebuhr J, Weiss SR, Kalinke U, Thiel V. Early endonuclease-mediated evasion of RNA sensing ensures efficient coronavirus replication. PLoS Pathog. 2017 Feb 3;13(2):e1006195. doi: 10.1371/journal.ppat.1006195. eCollection 2017 Feb. PMID 28158275
- [Result] Kumaki Y, Salazar AM, Wandersee MK, Barnard DL. Prophylactic and therapeutic intranasal administration with an immunomodulator, Hiltonol(R) (Poly IC:LC), in a lethal SARS-CoV-infected BALB/c mouse model. Antiviral Res. 2017 Mar;139:1-12. doi: 10.1016/j.antiviral.2016.12.007. Epub 2016 Dec 9. PMID 27956136
- [Result] Longhi MP, Trumpfheller C, Idoyaga J, Caskey M, Matos I, Kluger C, Salazar AM, Colonna M, Steinman RM. Dendritic cells require a systemic type I interferon response to mature and induce CD4+ Th1 immunity with poly IC as adjuvant. J Exp Med. 2009 Jul 6;206(7):1589-602. doi: 10.1084/jem.20090247. Epub 2009 Jun 29. PMID 19564349
- [Result] Marcus PI, Sekellick MJ. Combined sequential treatment with interferon and dsRNA abrogates virus resistance to interferon action. J Interferon Cytokine Res. 2001 Jun;21(6):423-9. doi: 10.1089/107999001750277907. PMID 11440640
- [Result] Packard AE, Hedges JC, Bahjat FR, Stevens SL, Conlin MJ, Salazar AM, Stenzel-Poore MP. Poly-IC preconditioning protects against cerebral and renal ischemia-reperfusion injury. J Cereb Blood Flow Metab. 2012 Feb;32(2):242-7. doi: 10.1038/jcbfm.2011.160. Epub 2011 Nov 16. PMID 22086194
- [Result] Pavlick A, Blazquez AB, Meseck M, Lattanzi M, Ott PA, Marron TU, Holman RM, Mandeli J, Salazar AM, McClain CB, Gimenez G, Balan S, Gnjatic S, Sabado RL, Bhardwaj N. Combined Vaccination with NY-ESO-1 Protein, Poly-ICLC, and Montanide Improves Humoral and Cellular Immune Responses in Patients with High-Risk Melanoma. Cancer Immunol Res. 2020 Jan;8(1):70-80. doi: 10.1158/2326-6066.CIR-19-0545. Epub 2019 Nov 7. PMID 31699709
- [Result] Rockx B, Baas T, Zornetzer GA, Haagmans B, Sheahan T, Frieman M, Dyer MD, Teal TH, Proll S, van den Brand J, Baric R, Katze MG. Early upregulation of acute respiratory distress syndrome-associated cytokines promotes lethal disease in an aged-mouse model of severe acute respiratory syndrome coronavirus infection. J Virol. 2009 Jul;83(14):7062-74. doi: 10.1128/JVI.00127-09. Epub 2009 May 6. PMID 19420084
- [Result] Ruan Q, Yang K, Wang W, Jiang L, Song J. Clinical predictors of mortality due to COVID-19 based on an analysis of data of 150 patients from Wuhan, China. Intensive Care Med. 2020 May;46(5):846-848. doi: 10.1007/s00134-020-05991-x. Epub 2020 Mar 3. No abstract available. PMID 32125452
- [Result] Sabbatini P, Tsuji T, Ferran L, Ritter E, Sedrak C, Tuballes K, Jungbluth AA, Ritter G, Aghajanian C, Bell-McGuinn K, Hensley ML, Konner J, Tew W, Spriggs DR, Hoffman EW, Venhaus R, Pan L, Salazar AM, Diefenbach CM, Old LJ, Gnjatic S. Phase I trial of overlapping long peptides from a tumor self-antigen and poly-ICLC shows rapid induction of integrated immune response in ovarian cancer patients. Clin Cancer Res. 2012 Dec 1;18(23):6497-508. doi: 10.1158/1078-0432.CCR-12-2189. Epub 2012 Oct 2. PMID 23032745
- [Result] Salazar AM, Levy HB, Ondra S, Kende M, Scherokman B, Brown D, Mena H, Martin N, Schwab K, Donovan D, Dougherty D, Pulliam M, Ippolito M, Graves M, Brown H, Ommaya A. Long-term treatment of malignant gliomas with intramuscularly administered polyinosinic-polycytidylic acid stabilized with polylysine and carboxymethylcellulose: an open pilot study. Neurosurgery. 1996 Jun;38(6):1096-103; discussion 1103-4. PMID 8727138
- [Result] Sultan H, Wu J, Kumai T, Salazar AM, Celis E. Role of MDA5 and interferon-I in dendritic cells for T cell expansion by anti-tumor peptide vaccines in mice. Cancer Immunol Immunother. 2018 Jul;67(7):1091-1103. doi: 10.1007/s00262-018-2164-6. Epub 2018 Apr 25. PMID 29696308
- [Result] Walberg K, Baron S, Poast J, Schwartz B, Izotova L, Pestka S, Peterson JW. Interferon protects mice against inhalation anthrax. J Interferon Cytokine Res. 2008 Oct;28(10):597-601. doi: 10.1089/jir.2007.0143. PMID 18778201
- [Result] Wang Y, Wang Y, Chen Y, Qin Q. Unique epidemiological and clinical features of the emerging 2019 novel coronavirus pneumonia (COVID-19) implicate special control measures. J Med Virol. 2020 Jun;92(6):568-576. doi: 10.1002/jmv.25748. Epub 2020 Mar 29. PMID 32134116
- [Result] Wong JP, Christopher ME, Viswanathan S, Dai X, Salazar AM, Sun LQ, Wang M. Antiviral role of toll-like receptor-3 agonists against seasonal and avian influenza viruses. Curr Pharm Des. 2009;15(11):1269-74. doi: 10.2174/138161209787846775. PMID 19355966
- [Result] Wong JP, Saravolac EG, Sabuda D, Levy HB, Kende M. Prophylactic and therapeutic efficacies of poly(IC.LC) against respiratory influenza A virus infection in mice. Antimicrob Agents Chemother. 1995 Nov;39(11):2574-6. doi: 10.1128/AAC.39.11.2574. PMID 8585749
- [Result] Zhou Q, Chen V, Shannon CP, Wei XS, Xiang X, Wang X, Wang ZH, Tebbutt SJ, Kollmann TR, Fish EN. Interferon-alpha2b Treatment for COVID-19. Front Immunol. 2020 May 15;11:1061. doi: 10.3389/fimmu.2020.01061. eCollection 2020. PMID 32574262
- [Result] Zhu X, Fallert-Junecko BA, Fujita M, Ueda R, Kohanbash G, Kastenhuber ER, McDonald HA, Liu Y, Kalinski P, Reinhart TA, Salazar AM, Okada H. Poly-ICLC promotes the infiltration of effector T cells into intracranial gliomas via induction of CXCL10 in IFN-alpha and IFN-gamma dependent manners. Cancer Immunol Immunother. 2010 Sep;59(9):1401-9. doi: 10.1007/s00262-010-0876-3. Epub 2010 Jun 12. PMID 20549206
- [Result] Field AK, Tytell AA, Piperno E, Lampson GP, Nemes MM, Hilleman MR. Poly I:C, an inducer of interferon and interference against virus infections. Medicine (Baltimore). 1972 May;51(3):169-74. doi: 10.1097/00005792-197205000-00002. No abstract available. PMID 4336643
- [Result] Gesuete R, Christensen SN, Bahjat FR, Packard AE, Stevens SL, Liu M, Salazar AM, Stenzel-Poore MP. Cytosolic Receptor Melanoma Differentiation-Associated Protein 5 Mediates Preconditioning-Induced Neuroprotection Against Cerebral Ischemic Injury. Stroke. 2016 Jan;47(1):262-6. doi: 10.1161/STROKEAHA.115.010329. Epub 2015 Nov 12. PMID 26564103
- [Result] Harrington DG, Crabbs CL, Hilmas DE, Brown JR, Higbee GA, Cole FE Jr, Levy HB. Adjuvant effects of low doses of a nuclease-resistant derivative of polyinosinic acid . polycytidylic acid on antibody responses of monkeys to inactivated Venezuelan equine encephalomyelitis virus vaccine. Infect Immun. 1979 Apr;24(1):160-6. doi: 10.1128/iai.24.1.160-166.1979. PMID 110688
- [Result] Ivanova A, Qaqish BF, Schell MJ. Continuous toxicity monitoring in phase II trials in oncology. Biometrics. 2005 Jun;61(2):540-5. doi: 10.1111/j.1541-0420.2005.00311.x. PMID 16011702
- [Result] Levine AS, Sivulich M, Wiernik PH, Levy HB. Initial clinical trials in cancer patients of polyriboinosinic-polyribocytidylic acid stabilized with poly-L-lysine, in carboxymethylcellulose [poly(ICLC)], a highly effective interferon inducer. Cancer Res. 1979 May;39(5):1645-50. No abstract available. PMID 371793
- [Result] Martins KAO, Cooper CL, Stronsky SM, Norris SLW, Kwilas SA, Steffens JT, Benko JG, van Tongeren SA, Bavari S. Adjuvant-enhanced CD4 T Cell Responses are Critical to Durable Vaccine Immunity. EBioMedicine. 2015 Nov 27;3:67-78. doi: 10.1016/j.ebiom.2015.11.041. eCollection 2016 Jan. PMID 26870818
- [Result] Okada H, Butterfield LH, Hamilton RL, Hoji A, Sakaki M, Ahn BJ, Kohanbash G, Drappatz J, Engh J, Amankulor N, Lively MO, Chan MD, Salazar AM, Shaw EG, Potter DM, Lieberman FS. Induction of robust type-I CD8+ T-cell responses in WHO grade 2 low-grade glioma patients receiving peptide-based vaccines in combination with poly-ICLC. Clin Cancer Res. 2015 Jan 15;21(2):286-94. doi: 10.1158/1078-0432.CCR-14-1790. Epub 2014 Nov 25. PMID 25424847
- [Result] Rosenfeld MR, Chamberlain MC, Grossman SA, Peereboom DM, Lesser GJ, Batchelor TT, Desideri S, Salazar AM, Ye X. A multi-institution phase II study of poly-ICLC and radiotherapy with concurrent and adjuvant temozolomide in adults with newly diagnosed glioblastoma. Neuro Oncol. 2010 Oct;12(10):1071-7. doi: 10.1093/neuonc/noq071. Epub 2010 Jul 8. PMID 20615924
- [Result] Sahin U, Muik A, Derhovanessian E, Vogler I, Kranz LM, Vormehr M, Baum A, Pascal K, Quandt J, Maurus D, Brachtendorf S, Lorks V, Sikorski J, Hilker R, Becker D, Eller AK, Grutzner J, Boesler C, Rosenbaum C, Kuhnle MC, Luxemburger U, Kemmer-Bruck A, Langer D, Bexon M, Bolte S, Kariko K, Palanche T, Fischer B, Schultz A, Shi PY, Fontes-Garfias C, Perez JL, Swanson KA, Loschko J, Scully IL, Cutler M, Kalina W, Kyratsous CA, Cooper D, Dormitzer PR, Jansen KU, Tureci O. COVID-19 vaccine BNT162b1 elicits human antibody and TH1 T cell responses. Nature. 2020 Oct;586(7830):594-599. doi: 10.1038/s41586-020-2814-7. Epub 2020 Sep 30. PMID 32998157
- [Result] Stephen EL, Hilmas DE, Mangiafico JA, Levy HB. Swine influenza virus vaccine: potentiation of antibody responses in rhesus monkeys. Science. 1977 Sep 23;197(4310):1289-90. doi: 10.1126/science.408923.
- [Result] Food and Drug Administration, HHS. International Conference on Harmonisation; Guidance on E7 Studies in Support of Special Populations; Geriatrics; Questions and Answers; availability. Notice. Fed Regist. 2012 Feb 21;77(34):9948-9. PMID 22379685